CLINICAL TRIAL: NCT07256743
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Determine the Efficacy SALI-10 Oral Probiotics in Experimental Gingivitis
Brief Title: Efficacy of SALI-10 Oral Probiotics in Experimental Gingivitis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ostia Sciences (Industry)
Collaborators: University of Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: OstiaGingivitis
Record Dates: First submitted 2025-09-23; First posted 2025-12-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-09

CONDITIONS: Gingivitis
Keywords: Probiotic; Oral Health; Lozenge
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Intervention Model Description: Once a participant volunteers they begin with a baseline visit. They receive a full oral assessment (probing depth, attachment level, plaque, gingival and bleeding indices) and biospecimen collection (gingival crevicular fluid, plaque, saliva, rinse); and is then assigned a study product: two lozenges (either active or placebo) daily for 14 days, taken after brushing, with instructions to maintain hygiene and return lozenge containers for compliance.
  Participants attend eight visits. At each, containers are returned, oral exams repeated, biospecimens collected, and questionnaires completed on product use and adverse events. During the induction phase (Day 0-21), subjects refrain from oral hygiene while continuing lozenges twice daily. On Day 21, participants receive prophylaxis and resume oral hygiene while continuing lozenges for two weeks.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (No Intervention): Placebo lozenges used
- SALI-10 (Active Comparator): Lozenges containing 6B CFUs of
  Interventions: Dietary Supplement: 6B SALI-10

INTERVENTIONS:
Dietary Supplement: 6B SALI-10 — Lozenges containing 6B CFUs of probiotic S. salivarius SALI-10
  Arms: SALI-10

SUMMARY:
Gingivitis is among the most prevalent oral diseases worldwide, affecting an estimated 50-90% of adults. It is a reversible condition primarily caused by microbial plaque accumulation on teeth and gingival surfaces, which triggers inflammation. Standard care emphasizes plaque reduction through oral hygiene, and research shows gingivitis can be reversed once hygiene resumes. The classic experimental gingivitis (EG) model developed in 1965 by Löe and Silness demonstrated the direct link between plaque buildup and gingival inflammation, further confirming that gingival health can be restored after resuming proper care.

Microbial ecology shifts are central to gingivitis pathogenesis. In health, the oral microbiome is dominated by gram-positive Streptococcus species. With plaque accumulation, microbial communities transition to gram-negative periopathogens such as Porphyromonas, Tannerella, Treponema, and Prevotella. This dysbiosis provokes heightened inflammation, tissue damage, and, in susceptible individuals, progression to periodontitis. Individual variability in the inflammatory response has been associated with differences in the presence and activity of beneficial streptococci. Certain strains of Streptococcus salivarius produce lantibiotics called salivaricins-polycyclic antimicrobial peptides containing lanthionine residues. Salivaricins inhibit oral pathogens and have been investigated for their antimicrobial and probiotic properties, particularly in the context of rising antibiotic resistance. Probiotic S. salivarius strains isolated from healthy individuals have demonstrated safety and antimicrobial potential in previous studies, supporting their use in preventing oral and respiratory infections.

A strain of S. salivarius designated SALI-10 produces a lantibiotic, Salivaricin 10, and is being evaluated as a candidate for gingivitis prevention. This strain is hypothesized to (1) help stabilize populations of beneficial streptococci during plaque accumulation, (2) competitively inhibit periopathogens such as Porphyromonas and Prevotella, and (3) suppress the dysbiotic shift toward gram-negative dominance. By contributing to microbial balance and reducing inflammatory triggers, SALI-10 may support resilient host-microbe interactions associated with gingival health. This approach may offer a dual antimicrobial and microbiome-stabilizing strategy with relevance to gingivitis management and longer-term periodontal health.

DETAILED DESCRIPTION:
Gingivitis is an oral disease condition affecting 50% to 90% of adults globally. The gingivitis pathology can be reversed by reduction or removal of microbial plaque that accumulates on hard and soft tissues and is considered standard of care in the industry. Regular oral hygiene in combination with therapeutics that delivers an anti-microbial benefit is thought to mitigate the onset of gingivitis. However, testing therapeutics for prophylaxis benefit to mitigate development of gingivitis has not been fully examined.

The classical model of experimental gingivitis (EG) was developed in 1965 by Loe and Silness who convincingly demonstrated the causative relationship between the accumulation of dental plaque and the development of clinically evident gingivitis in healthy young adults abstaining from all oral hygiene practices for a 21-day period. Furthermore, on resuming customary oral hygiene practices, all subjects demonstrated a return to gingival health. Understanding how participants returned quickly to gingival health aligns with the current understanding that the clinically healthy state is an active and dynamic process.

Neutrophils, a type of white blood cell (leukocyte), represent a key component of the innate defence system that protects periodontal tissue from both gingivitis and periodontitis. Not only are they the first line of cellular defence, but they are among the most abundant leukocytes within the periodontal tissues. Gingivitis is associated with a significant increase in the number of neutrophils that migrate to periodontal tissue. In contrast, individuals with too few neutrophils brought about by either congenital deficiencies in neutrophil numbers or transit (LAD 1 and 2), or those with induced neutropenia by chemical induction with antimitotic agents such as cyclophosphamide, invariably develop periodontitis. Likewise, studies in knockout mice that are defective in neutrophil transit also develop periodontitis. Consistent with the key contribution of neutrophils to both gingivitis and periodontitis, neutrophil transit to gingival tissue is highly regulated. The periodontium contains innate host defense mediators that facilitate the transit of neutrophils from the highly vascularized gingival tissue to the gingival crevice, where they form a "wall" between the host tissue and the dental plaque biofilm.

However, the prolonged presence of neutrophils in gingival tissue is not tolerated in the healthy state. The failure to downregulate neutrophil transit results in an increase in neutrophil numbers in gingival tissue and a significant increase in periodontal bone loss. Therefore, neutrophil homing to the gingival crevice is highly regulated such that under conditions of periodontal health the appropriate amount of neutrophils are present to maintain control of dental plaque bacterial growth and yet not elicit tissue damage. Evaluation of oral and blood neutrophils during experimental gingivitis has shown that people with uniquely high inflammatory response have an exaggerated polymorphonuclear neutrophil response both in the oral cavity and in the blood.

Gingivitis is a reversible inflammatory condition caused by the accumulation of dental plaque and the associated disruption of the host-microbial homeostasis. During gingivitis, the microbial community transitions from being dominated by gram-positive health-associated bacteria, such as Streptococcus species, to gram-negative periopathogens, including species of the genera Porphyromonas, Tannerella, Treponema and Prevotella. This dysbiotic shift triggers inflammatory responses, leading to tissue damage and, in some cases, progression to periodontitis.

A recent study on human experimental gingivitis identified three distinct host response phenotypes-high, low, and slow responders-based on clinical, inflammatory, and microbial parameters:

High Responders: Rapid plaque accumulation accompanied by a significant increase in gram-negative periopathogens and elevated inflammatory markers, such as interleukin-1β (IL-1β).

Low Responders: Similar plaque accumulation to high responders but lower inflammation, suggesting a more muted host response to bacterial dysbiosis.

Slow Responders: Delayed plaque accumulation and microbial succession, with prolonged dominance of health-associated Streptococcus species and a delayed or reduced inflammatory response.

Microbial analysis revealed that the persistence of beneficial Streptococcus species, such as S. sanguinis and S. oralis, in slow and low responders correlates with a protective effect against the emergence of periopathogens and the associated inflammatory cascade. Conversely, the loss of these beneficial bacteria in high responders was linked to more severe inflammation, highlighting the critical role of the oral microbiome in modulating gingivitis severity.

Lantibiotic salivaricins are polycyclic peptides containing lanthionine and/or β-methyllanthionine residues that are produced by certain strains of Streptococcus salivarius, which almost exclusively reside in the human oral cavity. These molecules are notable for their antimicrobial activity toward relevant oral pathogens, supporting the development of salivaricin-producing probiotic strains. Salivaricins are also relevant for development of novel antibacterial therapies in the context of emerging antibiotic resistance. Previous work has shown the bacteriocin and safety features of S. salivarius strains isolated from healthy subjects, demonstrating their potential for use as probiotics.

Proposed Solution: S. salivarius SALI-10

The investigators propose using a novel strain, Streptococcus salivarius SALI-10, as a targeted microbial intervention to modulate the oral microbiome and prevent gingivitis. S. salivarius SALI-10 is hypothesized to:

* Maintain a stable population of beneficial streptococci during plaque accumulation.
* Inhibit the growth of periopathogens through microbial competition and production of Salivaricin 10.
* Delay or suppress the dysbiotic shift to gram-negative dominance, thereby reducing the inflammatory response.

By supporting microbial homeostasis, SALI-10 may emulate the resilience observed in slow responders and offer a novel strategy for gingivitis prevention.

Dosage Regimen

This is a placebo-controlled study. Each participant randomized to the intervention group will receive mint-flavoured SALI-10 lozenges. They will take one lozenge twice a day-morning and evening-after brushing, allowing it to dissolve in the mouth. Participants will use the study lozenges throughout the study.

Prestudy Screening and Baseline Evaluation Telephone Pre-Screening

Potential study participants who express interest will be contacted by telephone. Eligibility for screening will be assessed using standard recruitment questions.

In-Person Screening

Before screening procedures occur, participants will provide informed consent. Participants will complete demographic and health information and undergo an oral examination of soft and hard tissues. Female participants will undergo a urine pregnancy test. The screening continues until sixty (60) participants are enrolled.

Visit 1 - Baseline Assessment

Participants will undergo an oral exam including probing depth (PD), attachment level (AL), visible plaque index (VPI), gingival index (GI), and bleeding on probing (BOP). Biospecimens collected will include gingival crevicular fluid (GCF), subgingival plaque, saliva, and an oral rinse. Participants will receive a dental cleaning and their assigned study product with instructions.

Treatment Visit Schedule

Participants will consume two lozenges per day at home and attend eight (8) study visits.

Visit 2 (Day -14 / -7)

Oral examination and biospecimen collection (GCF, plaque, saliva, oral rinse). Participants report use of NHPs and adverse effects.

Induction Phase (No Oral Hygiene for 21 Days) Visit 3 (Day 0)

Oral examination and biospecimen collection. Participants refrain from all oral hygiene for 21 days and continue their assigned lozenges.

Visit 4 (Day 7)

Oral examination and biospecimen collection. Participants are reminded to continue refraining from oral hygiene.

Visit 5 (Day 14)

Oral examination and biospecimen collection. Participants continue refraining from oral hygiene.

Resolution Phase (Participants Resume Oral Hygiene) Visit 6 (Day 21)

Oral examination and biospecimen collection. Participants receive a dental cleaning and resume home oral hygiene while continuing study lozenges.

Visit 7 (Day 28)

Oral examination and biospecimen collection.

Visit 8 - End of Study (Day 35)

Oral examination and biospecimen collection. Participants receive compensation and resume regular oral hygiene. After study completion, the manufacturer will unblind the product groups, and participants will be informed of their assignment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female volunteers aged 18-70 years
2. In good general health, ASA I
3. No clinical signs of gingival inflammation at >90% of sites observed
4. Absence of Periodontal Pockets, Probing Depth (PD) < 3.0 mm on all teeth/site
5. Absence of Clinical Attachment Loss (CAL) = 0 mm
6. No periodontal disease history
7. Have at least 20 gradeable teeth
8. Non-smokers
9. Fluent in English
10. For study participants of childbearing potential, both men and women, at least one of the following birth control measures must be used: abstinence, hormonal birth control (oral, injectable, transdermal, intra-vaginal), intrauterine devices, confirmed successful vasectomy, or condoms.

Exclusion Criteria:

1. Presence of orthodontic bands.
2. Presence of partial or full dentures.
3. Tumour(s) of the soft or the hard tissues of the oral cavity.
4. Cavitated carious lesions requiring immediate restorative treatment.
5. History of allergy to a consumer or personal care products or dentifrice ingredients as determined by the dental profession monitoring the study.
6. Participation in any other clinical study or test panel within one month before entering the study.
7. Medical condition which requires pre-medication before dental visits/procedures
8. Current use of anti-inflammatory, antibiotics, or antimicrobial drugs or within the last 30 days of enrolment.
9. History of periodontal disease.
10. History of systemic inflammatory, immune conditions and immunocompromised conditions
11. Pregnant or nursing women or those planning to get pregnant
12. Use of tobacco products.
13. Long-term antibiotic or anti-inflammatory therapy.
14. Medication or Natural Health Products (NHPs) that could affect the gingiva like calcium channel blockers, anti-epileptic therapy etc.
15. Medical condition or any current usage of medication that the investigator considers may compromise the study participant's safety as well as the quality of the study results
16. Allergy to any of the following ingredients: Streptococcus Salivarius, Sorbitol, Isomalt, Calcium phosphate dibasic, Potato starch, Mint, Glyceryl dibehenate, Stevia, Maltodextrin
17. Use of other probiotics
18. Taking anticoagulant medications and those suffering from blood and bleeding disorders
19. Recently experienced or will be experiencing dental, oral or any type of surgery.
20. Use of anti-plaque/ anti-gingivitis products
21. Presence of active infections
22. Participants who are experiencing nausea, fever, vomiting, bloody diarrhoea or severe abdominal pain.
23. Use of any antibiotics.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Mean change in percentage of sites with bleeding on probing (BOP) | Baseline; Weeks 1 and 2 (pre-induction); Weeks 3 - 5 (induction phase - no-brushing); Weeks 6 and 7 (resolution phase).
  Bleeding on probing (BOP) will be assessed at six sites per tooth using a UNC-15 periodontal probe. The proportion of bleeding sites (% of total sites) will be calculated for each participant. Group mean ± SD change from baseline will be reported.
  Scale: 0-100 %; lower values = less gingival inflammation.

SECONDARY OUTCOMES:
Change in oral neutrophil (oPMN) count per 10 mL unstimulated saliva | Baseline; Weeks 1 and 2 (pre-induction); Weeks 3 - 5 (induction phase - no-brushing); Weeks 6 and 7 (resolution phase).
  Unstimulated saliva (10 mL) will be collected, centrifuged, and stained with acridine orange. Neutrophils will be counted using fluorescence microscopy and a hemocytometer. Results expressed as total PMNs × 10³ cells / 10 mL.
Change in concentration of cytokines (IL-1β, IL-6, MMP-8) in gingival crevicular fluid (pg/mL) | Baseline; Weeks 1 and 2 (pre-induction); Weeks 3 - 5 (induction phase - no-brushing); Weeks 6 and 7 (resolution phase).
  Gingival crevicular fluid (GCF) will be collected using Periopaper strips and analyzed with bead-based multiplex immunoassays (Luminex). Mean concentrations (pg/mL) will be reported per participant; lower values indicate reduced local inflammation.
Change in relative abundance of periodontal and commensal bacteria measured by quantitative PCR and shotgun metagenomics | Baseline; Weeks 1 and 2 (pre-induction); Weeks 3 - 5 (induction phase - no-brushing); Weeks 6 and 7 (resolution phase).
  DNA extracted from subgingival plaque and tongue swabs will be analyzed for P. gingivalis, F. nucleatum, T. forsythia, P. micra and S. salivarius SALI-10. Abundance expressed as ΔCt relative to total 16S rRNA gene copies. Metagenomic analysis will evaluate community shifts.
Change in concentration of volatile sulfur compounds (VSCs) in exhaled air measured by Halimeter (ppb) | Baseline; Weeks 1 and 2 (pre-induction); Weeks 3 - 5 (induction phase - no-brushing); Weeks 6 and 7 (resolution phase).
  Halitosis will be quantified using a calibrated Halimeter (Interscan Corp.). Three consecutive breath readings will be averaged per visit. Results reported in parts per billion (ppb); lower values indicate improved oral odor.
Change in mean Gingival Index (GI) score | Baseline; Weeks 1 and 2 (pre-induction); Weeks 3 - 5 (induction phase - no-brushing); Weeks 6 and 7 (resolution phase).
  Gingival inflammation will be assessed using the Löe-Silness Gingival Index. Scale: 0 = normal; 1 = mild; 2 = moderate; 3 = severe. Lower mean scores indicate improved gingival health.
Change in mean Plaque Index (PI) score | Baseline; Weeks 1 and 2 (pre-induction); Weeks 3 - 5 (induction phase - no-brushing); Weeks 6 and 7 (resolution phase).
  Plaque accumulation will be assessed using the Silness-Löe Plaque Index. Scale: 0 = no plaque; 1 = thin film; 2 = moderate deposits; 3 = abundant plaque.
  Lower mean scores indicate improved oral hygiene.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Michael Goldberg, MDM, Principal Investigator — University of Toronto
Locations (1):
- University of Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
No individual participant data (IPD) will be shared. IPD will not be shared because the data include proprietary early-stage clinical development information that is not intended for public release.

REFERENCES:
- [Background] Wellappuli NC, Fine N, Lawrence HP, Goldberg M, Tenenbaum HC, Glogauer M. Oral and Blood Neutrophil Activation States during Experimental Gingivitis. JDR Clin Trans Res. 2018 Jan;3(1):65-75. doi: 10.1177/2380084417742120. Epub 2017 Nov 20. PMID 30938653
- [Background] van der Weijden F, Slot DE. Oral hygiene in the prevention of periodontal diseases: the evidence. Periodontol 2000. 2011 Feb;55(1):104-23. doi: 10.1111/j.1600-0757.2009.00337.x. No abstract available. PMID 21134231
- [Background] LOE H, THEILADE E, JENSEN SB. EXPERIMENTAL GINGIVITIS IN MAN. J Periodontol (1930). 1965 May-Jun;36:177-87. doi: 10.1902/jop.1965.36.3.177. No abstract available. PMID 14296927
- [Background] Kerns KA, Bamashmous S, Hendrickson EL, Kotsakis GA, Leroux BG, Daubert DD, Roberts FA, Chen D, Trivedi HM, Darveau RP, McLean JS. Localized microbially induced inflammation influences distant healthy tissues in the human oral cavity. Proc Natl Acad Sci U S A. 2023 Oct 10;120(41):e2306020120. doi: 10.1073/pnas.2306020120. Epub 2023 Oct 2. PMID 37782795
- [Background] Gunsolley JC. A meta-analysis of six-month studies of antiplaque and antigingivitis agents. J Am Dent Assoc. 2006 Dec;137(12):1649-57. doi: 10.14219/jada.archive.2006.0110. PMID 17138709
- [Background] Gallagher H, Ramsay SC, Barnes J, Maggs J, Cassidy N, Ketheesan N. Neutrophil labeling with [(99m)Tc]-technetium stannous colloid is complement receptor 3-mediated and increases the neutrophil priming response to lipopolysaccharide. Nucl Med Biol. 2006 Apr;33(3):433-9. doi: 10.1016/j.nucmedbio.2005.12.014. Epub 2006 Mar 9. PMID 16631093
- [Background] Berezow AB, Darveau RP. Microbial shift and periodontitis. Periodontol 2000. 2011 Feb;55(1):36-47. doi: 10.1111/j.1600-0757.2010.00350.x. No abstract available. PMID 21134227
- [Background] Barbour A, Wescombe P, Smith L. Evolution of Lantibiotic Salivaricins: New Weapons to Fight Infectious Diseases. Trends Microbiol. 2020 Jul;28(7):578-593. doi: 10.1016/j.tim.2020.03.001. Epub 2020 Apr 6. PMID 32544444
- [Background] Barbour A, Philip K. Variable characteristics of bacteriocin-producing Streptococcus salivarius strains isolated from Malaysian subjects. PLoS One. 2014 Jun 18;9(6):e100541. doi: 10.1371/journal.pone.0100541. eCollection 2014. PMID 24941127
- [Background] Albandar JM, Rams TE. Global epidemiology of periodontal diseases: an overview. Periodontol 2000. 2002;29:7-10. doi: 10.1034/j.1600-0757.2002.290101.x. No abstract available. PMID 12102700

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2025-10-11): https://cdn.clinicaltrials.gov/large-docs/43/NCT07256743/Prot_ICF_000.pdf